CLINICAL TRIAL: NCT06478069
Title: Postural Assessment of Stroke Patients by Pose Estimation and Effects of Dynamic Core Postural Chain Stabilization Techniques
Brief Title: Postural Assessment of Stroke Patients by Pose Estimation and Effects of Dynamic Core Postural Chain Stabilization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/722
Record Dates: First submitted 2024-06-10; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Chromosomes, Human, 1-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other)
  Interventions: Diagnostic Test: Group A
- Group B (Experimental)
  Interventions: Behavioral: Group B

INTERVENTIONS:
Diagnostic Test: Group A — Group A was treated with Ibuprofen Dosage After breakfast and after dinner for 6 weeks.
  Arms: Group A
Behavioral: Group B — Group B was treated with physical therapy; (Upper limb: The stroke patient warmed up with some gentle stretches for the wrist and fingers to get the muscles ready. They subsequently engaged in resistance training using dumbbells or resistance bands to increase the strength of their upper limbs. Bicep curls, tricep extensions, and shoulder presses were some of these exercises. They tried to complete two to three sets of ten to fifteen repetitions for each exercise, progressively increasing the resistance as their strength increased. Then, to improve dexterity and coordination in daily tasks, functional exercises were included.
  Arms: Group B

SUMMARY:
This study focuses on a two-pronged strategy to enhance the rehabilitation of stroke patients. It first investigates the application of pose estimating technologies to objectively measure posture.

DETAILED DESCRIPTION:
This can entail capturing a patient's body position with cameras or other sensors in order to detect any imbalances or variations from normal posture brought on by the stroke. The study also looks at how well dynamic core postural chain stabilization (DCS) methods work for stroke recovery. The goal of DCS exercises is to increase stability and strength in the core, which can help with general postural control. This research aims to optimize stroke patient rehabilitation by combining a precise evaluation approach with a focused intervention strategy, which may result in improved balance, movement, and functional abilities.

ELIGIBILITY:
Inclusion Criteria:

* Stroke, either ischemic or hemorrhagic
* Standing ability and ability to perform basic movements with assistance
* Willingness to take part in the intervention and evaluations

Exclusion Criteria:

* Severe cognitive impairment hindering participation
* Unstable medical conditions affecting rehabilitation
* History of other neurological disorders affecting posture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 12 Months
  For evaluating balance in a variety of functional tasks, the BBS is a commonly used and validated test. After the intervention period, the BBS scores of the control group and the intervention group (who received DCS techniques) can be compared. The efficacy of DCS in enhancing postural control would be strongly supported by a statistically significant increase in the intervention group's BBS score.
Trunk Impairment Scale (TIS) Score | 12 months
  The total score for TIS ranges between 0 for a minimal performance to 23 for a perfect performance. In a recent version of the TIS (version 2.0) for adults, the static subscale was removed because of a ceiling effect, total score ranges between 0 and 16 points

CONTACTS AND LOCATIONS:
Locations (1):
- Sevices Hospital Shadman 1, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No